CLINICAL TRIAL: NCT01613066
Title: Intra-bone Cord Blood Transplantation in Patients With Haematological Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, Roberto Sorasio, MD, Ospedale Santa Croce-Carle Cuneo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Emato68
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: High Risk Haematological Malignancies; Advanced Haematological Malignancies
Keywords: Haematological malignancies; Allogeneic Cord Blood transplantation; Intrabone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients with high risk haematological malignancies
  Interventions: Procedure: Intrabone Allogeneic Transplant

INTERVENTIONS:
Procedure: Intrabone Allogeneic Transplant — Unrelated single unit intrabone cord blood transplantation

SUMMARY:
Cord blood (CB) from an unrelated donor is increasingly used an alternative source of hematopoietic stem cells for adults with hematologic malignancies who lack an HLA-matched donor. However, the utilization of single-unit CB for transplantation of adult patients has been impeded by the low number of nucleated cells available from individual CB units. Direct intrabone CB injection (IBCBi) has been recently investigated as a solution to cell dose problem in adults, with the aims of minimizing non-specific loss of progenitors. We set up a phase I-II study to assess the safety and efficacy of CB transplantation by IBCBi in adult patients with advanced or high-risk hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

* Advanced or High Risk Haematological Malignancies
* Age 18-65 years
* no suitable unrelated HLA-matched donors identified in a clinically useful time-frame
* Informed consent

Exclusion Criteria:

* Active infectious disease at inclusion
* HIV- positivity or active hepatitis infection
* Impaired liver function (Bilirubin > upper normal limit; Transaminases > 3.0 x upper normal limit) at inclusion
* Impaired renal function (Creatinine-clearance <60 ml/min; Serum Creatinine >1.5 x upper normal limit) at inclusion
* Psychiatric diseases or conditions that might impair the ability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Time to neutrophil recovery | 28 days after transplantation

SECONDARY OUTCOMES:
Incidence of platelet engraftment | 100 days after transplantation
Acute graft versus host disease | 100 days after transplantation
Chronic Graft Versus Host Disease | One year after transplantation
Overall Survival | One year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Mattei, MD, Principal Investigator — ASO S Croce e Carle
Locations (1):
- Azienda Ospedaliera S Croce e Carle, Cuneo, Cuneo, Italy

REFERENCES:
- [Background] Frassoni F, Gualandi F, Podesta M, Raiola AM, Ibatici A, Piaggio G, Sessarego M, Sessarego N, Gobbi M, Sacchi N, Labopin M, Bacigalupo A. Direct intrabone transplant of unrelated cord-blood cells in acute leukaemia: a phase I/II study. Lancet Oncol. 2008 Sep;9(9):831-9. doi: 10.1016/S1470-2045(08)70180-3. Epub 2008 Aug 8. PMID 18693069
- [Background] Page KM, Zhang L, Mendizabal A, Wease S, Carter S, Gentry T, Balber AE, Kurtzberg J. Total colony-forming units are a strong, independent predictor of neutrophil and platelet engraftment after unrelated umbilical cord blood transplantation: a single-center analysis of 435 cord blood transplants. Biol Blood Marrow Transplant. 2011 Sep;17(9):1362-74. doi: 10.1016/j.bbmt.2011.01.011. Epub 2011 Jan 28. PMID 21277377